CLINICAL TRIAL: NCT03928470
Title: A Multicenter, Randomized, Double-blind, Active-controlled Phase 4 Study to Evaluate the Efficacy and Safety of EsoDuo Tab. 20/800mg in Patients With Non-erosive Reflux Disease(NERD)
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of EsoDuo Tab. 20/800mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 273GERD18019
Record Dates: First submitted 2019-04-15; First posted 2019-04-26 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Non-erosive Reflux Disease(NERD)
MeSH Terms: conditions — Non-Erosive Reflux Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EsoDuo Tab. 20/800mg (Experimental): EsoDuo Tab. 20/800mg
  Interventions: Drug: EsoDuo Tab. 20/800mg
- Nexium Tab. 20mg (Active Comparator): Nexium Tab. 20mg
  Interventions: Drug: EsoDuo Tab. 20/800mg

INTERVENTIONS:
Drug: EsoDuo Tab. 20/800mg — Nexium Tab. 20mg

SUMMARY:
To Evaluate the Efficacy and Safety of EsoDuo Tab. 20/800mg

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, active-controlled phase 4 study to evaluate the efficacy and safety of EsoDuo Tab. 20/800mg in patients with non-erosive reflux disease(NERD)

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female aged ≥ 19 years
2. Episode of heartburn for 3 months or more during prior to randomization visit.
3. Episode of heartburn for 2 days or more during the last 7 days prior to randomization visit.
4. Grade N, M by EGD test.

Exclusion Criteria:

1. Surgery history on stomach or esophagus
2. Active medical history of stomach, esophagus area
3. Other system disorder which can disturb this trial
4. Patients taking the contraindication of concomitant medications
5. Clinically significant Abnormal Lab test
6. Pregnant woman, Breastfeeding woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Complete resolution of heartburn(HB), Last 7 days of treatment, 4 weeks. | 4 weeks after drug administrations.
  Compare Experimental group with Active Comparator.

SECONDARY OUTCOMES:
Complete resolution of heartburn(HB), Last 7 days of treatment, 2 weeks. | 2 weeks after drug administrations
  Compare Experimental group with Active Comparator.
Complete resolution of Acid regurgitation, Last 7 days of treatment, 2 / 4 weeks. | 2/4 weeks after drug administrations.
  Compare Experimental group with Active Comparator.
The percentage of Heartburn(HB) / Acid regurgitation only 1 day or less free days, 2 / 4 weeks. | 2/4 weeks after drug administrations.
  Compare Experimental group with Active Comparator.
The percentage of free days without Heartburn(HB) / Acid regurgitation, 2 / 4 weeks. | 2/4 weeks after drug administrations.
  Compare Experimental group with Active Comparator.
The time to the first 24/48-h, 7-d of Heartburn(HB) / Acid regurgitation free interval. | 2/4 weeks after drug administrations.
  Compare Experimental group with Active Comparator.
Change from baseline in the Heartburn(HB) / Acid regurgitation Symptom score, 2 / 4 weeks. | 2/4 weeks after drug administrations.
  Compare Experimental group with Active Comparator.
Heartburn(HB) / Acid regurgitation symptoms per investigator assessment, 4weeks. | 4 weeks after drug administrations.
  Compare Experimental group with Active Comparator.
Time to first resolution of Heartburn(HB), Day 1 | 1 day after drug administrations.
  Compare Experimental group with Active Comparator.

CONTACTS AND LOCATIONS:
Overall Officials: Oh Young Lee, M.D., Ph.D., Principal Investigator — Hanyang University
Locations (38):
- South Korea (38):
  - Dong-A University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Chungbuk National University Hospital, Cheongju-si
  - Hallym University Chuncheon Seonsim Hospital, Chuncheon
  - Daegu Catholic Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medicar Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Myongji Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Ajou University Hospital, Gyeonggi-do
  - Hanyang University Guri Hospital, Gyeonggi-do
  - Inje University ilsan Paik Hospital, Gyeonggi-do
  - Soonchunhyang University Bucheon Hospital, Gyeonggi-do
  - Wonkwang University Hospital, Iksan
  - Dongguk University IIsan Hospital, Ilsan
  - Gachon Gil Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Chonbuk National University Hospital, Jeonju
  - Inje University Busan Paik Hospital, Pusan
  - Inje University Haeundae Paik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Yangsan Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul, Seoul
  - Catholic University Seoul St. Mary's Hospital, Seoul
  - Chung Ang University Hospital, Seoul
  - Gangnam Severance, Seoul
  - Hanyang University Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyunghee Universtiy Hospital, Seoul
  - Samsung Seoul Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SH, Lee KN, Lee OY, Choi MG, Kim JH, Sung IK, Jang JY, Park KS, Chun HJ, Kim EY, Lee JK, Jang JS, Kim GH, Hong SJ, Lee YC, Choi SC, Kim HS, Kim TO, Baik GH, Jeon YC. A Randomized, Double-Blind, Active-Control, Noninferiority, Multicenter, Phase 4 Study to Evaluate the Efficacy and Safety of Esomeprazole/Sodium Bicarbonate 20/800 mg in Patients with Nonerosive Gastroesophageal Reflux Disease. Gut Liver. 2023 Mar 15;17(2):226-233. doi: 10.5009/gnl220023. Epub 2022 Jun 22. PMID 35730245